CLINICAL TRIAL: NCT00361647
Title: Screening for Occult Malignancy in Idiopathic Venous Thromboembolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Paolo Prandoni, Department of Medical and Surgical Sciences, University of Padua
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 719P
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

INTERVENTIONS:
Procedure: Diagnostic screening for occult malignancy

SUMMARY:
Prospective controlled randomized study. Aim of this study is to assess the feasibility and sensitivity of CT scanning of the thorax, abdomen and pelvis for the detection of occult cancer in patients with idiopathic venous thromboembolism. Patients presenting with acute idiopathic venous thromboembolism, free from already known cancer and in whom a routine battery screening has excluded the presence of cancer, are randomized to receive either a CT scanning of the thorax, abdomen and pelvis (completed by mammography if not already performed in the past year, and by gastroscopy and/or colonoscopy in patients with positive hemoccult) or a diagnostic programme freely decided by attending physicians. Patients of either group in whom the search for cancer is negative are followed-up for two years to register the development of clinically symptomatic malignant disease. The rate of cancer detection and that of cancer development are compared between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic venous thromboembolism

Exclusion Criteria:

* cancer already known or shown by routine battery tests
* previous venous thromboembolism
* geographic inaccessibility for long-term follow-up
* allergy to contrast medium
* refusal of informed consensus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Prandoni, MD, PhD, Principal Investigator — Department of Medical and Surgical Sciences, University of Padua, Italy
Locations (1):
- Department of Medical and Surgical Sciences, 2nd Chair of Internal Medicine, University of Padua, Padua, Padua, Italy

REFERENCES:
- [Derived] Robertson L, Broderick C, Yeoh SE, Stansby G. Effect of testing for cancer on cancer- or venous thromboembolism (VTE)-related mortality and morbidity in people with unprovoked VTE. Cochrane Database Syst Rev. 2021 Oct 1;10(10):CD010837. doi: 10.1002/14651858.CD010837.pub5. PMID 34597414
- [Derived] Prandoni P, Bernardi E, Valle FD, Visona A, Tropeano PF, Bova C, Bucherini E, Islam MS, Piccioli A. Extensive Computed Tomography versus Limited Screening for Detection of Occult Cancer in Unprovoked Venous Thromboembolism: A Multicenter, Controlled, Randomized Clinical Trial. Semin Thromb Hemost. 2016 Nov;42(8):884-890. doi: 10.1055/s-0036-1592335. Epub 2016 Oct 20. PMID 27764880